CLINICAL TRIAL: NCT01912248
Title: Acute Effect of Strength Training on Blood Pressure in Cardiac Patients
Status: Completed | Type: Observational
Sponsor: Christian Dall (Other)
Responsible Party: Sponsor-Investigator, Christian Dall, cand.scient, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: H-2-2012-143
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure; Ischemic Heart Disease; Heart Transplant Recipients
Keywords: acute rise of systolic and diastolic bloodpressure
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Heart failure: strength training
  Interventions: Other: strength training
- Heart Transplant recipients: strength training
  Interventions: Other: strength training
- patients with ischemic heart disease: strength training
  Interventions: Other: strength training

INTERVENTIONS:
Other: strength training — strength training, lower limb.
  Other Names: one hour of strength training.

SUMMARY:
Moderate and heavy strength training exercise and the acute blood pressure rise in cardiac patient, how high?

DETAILED DESCRIPTION:
12 heart transplant recipients 12 heart failure patients 12 patients with ischemic heart disease

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* no strength training > 3 month
* speak and understand danish

Exclusion Criteria:

* cancer
* serum creatinin above 200 mmol/l
* re-transplantation
* Ejection fraction > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 12 heart transplant recipients 12 heart failure patients 12 patients with ischemic disease
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | one test, 1 hour, continuated systolic blood pressure surveliance

SECONDARY OUTCOMES:
diastolic blood pressure | one test 1 hour, continuated bloodpressure surveliance

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Dall, cand.scient, Principal Investigator — Bispebjerg Hospital, Denmark
Locations (1):
- Christian Dall, Copenhagen, Denmark